CLINICAL TRIAL: NCT07098312
Title: The Effect of Creative Drama Workshops Based on the Papadopoulos Model on the Cultural Competence Levels of Nursing Students: A Randomized Controlled Trial
Brief Title: Impact of Creative Drama on Nursing Students' Cultural Competence
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Yeter KITIS, Prof., Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: E-77082166-604.01-1204486
Record Dates: First submitted 2025-07-21; First posted 2025-08-01 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Cultural Competency
Keywords: creative drama; cultural competency; nursing students
MeSH Terms: interventions — Psychodrama

STUDY DESIGN:
Intervention Model Description: Randomized study with experimental and control groups
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the study, it is impossible to blind the researcher implementing the intervention and the participants. A pre-test will be administered before randomization to prevent bias in the study. The study's data collection and statistical process are planned to be blinded. The assignment of students to the intervention and control groups will be made by a statistician independent of the study. The researcher and the students will not know which group they are in until the application begins. After administering the follow-up tests, the independent researcher will code the data as groups A and B and transfer it to SPSS. With this method, the statistician plans to perform analysis and reporting without knowing which group is the intervention group and which is the control group. The codes of the groups are intended to be disclosed after the analysis and reporting of the data. In this way, detection bias, statistical bias, and reporting bias will be prevented.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Creative drama group (Experimental): Participants will be given eight sessions of creative drama intervention training in creative drama workshops reviewed by experts.
  Interventions: Behavioral: creative drama
- Control group (No Intervention): No intervention will be applied to the control group.

INTERVENTIONS:
Behavioral: creative drama — It is aimed to develop cultural competence in nursing students through creative drama workshops.
  Other Names: drama
  Arms: Creative drama group

SUMMARY:
The type of this research is a randomized controlled experimental study. The research aims to evaluate the effectiveness of creative drama workshops based on Papadopoulos' model on the cultural competence levels of nursing students. The population of the research consists of senior nursing students. The research sample will consist of at least 80 nursing students, 40 in the intervention group and 40 in the control group. The sample will be selected by randomization. 8 sessions of creative drama intervention will be applied to the students in the intervention group. The research aims to answer the following questions: Is there a difference between the intervention group and the control group in terms of cultural competence levels?

DETAILED DESCRIPTION:
With the impact of international migration, globalisation, and demographic changes, societies are becoming increasingly multicultural. The increase in cultural diversity poses a challenge to all social structures in any host country and also affects health care providers responsible for providing quality care to patients with diverse cultural backgrounds, especially those with health compliance needs In this context, working in a culturally diverse environment affects nurses the most as professionals who are directly interested in patient care and more closely experience cultural diversity. Providing culturally competent care places both a moral and a professional responsibility on nurses. Therefore, cultural competence education should have an important place in nursing programs whereby nursing students should be aware of their cultural values, beliefs, attitudes and behaviors and be able to communicate effectively with individuals with different cultural backgrounds In this direction, it is stated that the cultural competence trainings should be included in the nursing programs and intervention practices should be realized to improve the perceptions and skills of nursing students about their cultural care competencies.

Research with nursing students shows that levels of cultural competence are generally at an intermediate level. These studies suggest that interventions that improve cultural competence for nursing students are recommended. There are different theories, models or standards that guide interventions on cultural competence. One of them is the Papadopoulos Model.

Developed by Papadopoulos, Tilki and Taylor, the model is a continuous and successive model consisting of four dimensions of cultural awareness, cultural knowledge, cultural sensitivity and cultural practice to offer effective care in health care for the cultural beliefs and needs of individuals In the literature, there was no study using model-based and creative drama technique to increase cultural competence. Using creative drama, students try to understand how to integrate their theoretical knowledge into professional practice and explore how to react in various situations through a reflective process. Creative drama provides students with a clinical environment as close as possible to real life through players who portray patients, their relatives, and healthcare professionals. As a player or audience, students are involved in the evolving situation in real time and can imagine how they would react to it. They think about how they will react to these situations in a safe environment and can discuss these experiences with the instructor after observing the consequences of their decisions.

This project, which will be carried out to evaluate the effectiveness of creative drama workshops applied to nursing students based on the model of Papadopoulos, will use a randomized controlled experimental design by following the CONSORT guidelines.

Creative drama workshops will be applied to the intervention group. The creative drama workshops, which will be prepared based on the Papadopoulos model after the pre-testing, will be held in the practice laboratory of the Faculty of Nursing for two days a week for 4 weeks. To increase the effectiveness of creative drama applications, keeping the number of participants below 25 is important. This limitation is critical in increasing intra-group interaction, ensuring participants are more actively and efficiently involved. In this direction, the workshops are planned in two groups, each consisting of 20 people. Thus, both group dynamics will be maintained, and individual contributions of the participants will be allowed to come to the fore. These creative drama workshops aim to improve the cultural proficiency levels of nursing students, and in this process, they aim to increase cultural competence skills. Each workshop is planned to last two hours.

ELIGIBILITY:
Inclusion Criteria:

* Being a senior nursing student
* Participating in the study voluntarily
* Having a score below the average of the research population on the Cultural Competence Assessment Scale.

Exclusion Criteria:

* Having a diagnosed physical, mental, or psychological disorder
* Having previously received cultural competency training

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Cultural Competence Assessment Scale (CCAS) | six months
  The CCAS assesses cultural competence in four dimensions-cultural awareness, knowledge, sensitivity, and practice-each with 10 items. A total score is obtained by summing the scores from all sub-dimensions. If the score from cultural awareness is below 5, the person is classified as having "Cultural Inadequacy," regardless of other scores. A total score of 40 across all dimensions indicates "Cultural Competence." If the cultural awareness score is 5 or more and all of the first four items in the knowledge, sensitivity, and practice sub-dimensions are answered correctly, the level is defined as "Cultural Security." If the awareness score is 5 or more but there are incorrect answers among the first four items in the other sub-dimensions, the level is considered "Cultural Awareness."

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
IPD sharing is restricted by data confidentiality, participant privacy, and applicable ethics rules and legislation. Sharing data with third parties may require relevant ethics committee approval, institutional permissions, and explicit consent from participants. If these conditions are not met, IPD sharing may not be possible.